CLINICAL TRIAL: NCT01752959
Title: A Randomized Comparison of Esmolol and Remifentanil on Intraoperative Bleeding and Surgical Field Conditionsin Nasal Surgery
Brief Title: A Comparison of Esmolol and Remifentanil to Reduce Blood Loss
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Dondu Ruveyda Acikgoz, Medical Doctor Trainee in Anesthesiology and Reanimation, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RAcikgozEsmolol
Record Dates: First submitted 2012-12-04; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Deviation Septum Nasal
MeSH Terms: interventions — Remifentanil; esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanyl (Active Comparator): Group R 0.1-0.3 mic/kg/ min remifentanil infusion other names: Ultiva
  Interventions: Drug: Remifentanil
- esmolol (Experimental): Grup E 500 micg/kg/min lading dose after 50-500 μcg/kg/dk esmolol infusion
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Remifentanil — 0.1-0.3 micg/kg/min Remifentanil iv infusion
  Other Names: Ultiva
  Arms: Remifentanyl
Drug: Esmolol — 500 μcg/kg/dk esmolol iv lading dose after 50-500 μcg/kg/dk esmolol iv infusion
  Other Names: Brevibloc
  Arms: esmolol

SUMMARY:
In this prospective randomized study we aimed to compare the effects of esmolol and remifentanil on intraoperative bleeding surgical field conditions in nasal surgery

DETAILED DESCRIPTION:
60 patients with ASA I-IIphysical status assigned for septoplasty will be enrolled in this prospective randomized trial. A standardized anesthesia induction and intubation with propofol and rocuronium will be used. Patients will be randomized in two groups. Group Esmolol (Group E n=30) will receive esmolol 500 mic kg-1 loading dose and a 50-500 mic kg-1 min-1 infusion and Group Remifentanil (Group R n=30) will receive remifentanil 0.1-0.3 mic kg-1 min-1 infusion to induce controlled hypotension. A 50-60 mmHg mean arterial pressure and a minimum 50 beat min-1 heart rate is targeted. Heart rate, blood pressures, peripheral oxygen saturation and bispectral index spectrum (BIS) will be recorded. Anesthesia maintenance will be provided with O2/N2O and desflurane-propofol balanced anesthesia and a BIS value 40-60 is targeted. The quality of the surgical field will be assessed by the surgeon by using a 10 point visual analog scale (B1) and a 6 point scale (B2) during surgery with 5 minute intervals. The amount of bleeding will be calculated at the end of surgery from the amount of blood and irrigation fluid collected in the suction tube. All complications and side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II,
* between age 20-60

Exclusion Criteria:

* patients having bleeding disorders,
* arrhythmia,
* hypertension,
* endocrine, liver or kidney disease and
* those who are on antihypertensive,
* anticoagulant drugs

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the difference between group regarding blood loss | intraoperative
  controlled hypotension in nasal surgery

SECONDARY OUTCOMES:
the difference between groups regarding side effects and treatments | intraoperative
  side effects: more than 20% change in blood pressure and heart rate, treatment includes atropin, ephedrin, nitroglyserine

CONTACTS AND LOCATIONS:
Overall Officials: Ruveyda D Acıkgoz, Trainee, Principal Investigator — Ankara Diskapi Yildirim Beyazit Teaching and Research Hospital, Turkey.
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Degoute CS, Ray MJ, Manchon M, Dubreuil C, Banssillon V. Remifentanil and controlled hypotension; comparison with nitroprusside or esmolol during tympanoplasty. Can J Anaesth. 2001 Jan;48(1):20-7. doi: 10.1007/BF03019809. PMID 11212044
- [Background] Shen PH, Weitzel EK, Lai JT, Wormald PJ, Ho CS. Intravenous esmolol infusion improves surgical fields during sevoflurane-anesthetized endoscopic sinus surgery: a double-blind, randomized, placebo-controlled trial. Am J Rhinol Allergy. 2011 Nov-Dec;25(6):e208-11. doi: 10.2500/ajra.2011.25.3701. PMID 22185726